CLINICAL TRIAL: NCT01373957
Title: Long-tErm Follow-uP of Antithrombotic Management Patterns In Acute CORonary Syndrome Patients in RUSsia
Acronym: EPICOR-RUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CRU-XXX-2011/1
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; antithrombotic management; STEMI; NSTE-ACS
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients hospitalized and diagnosed with UA, STEMI or NSTEMI

SUMMARY:
EPICOR-RUS is a multi-centre, observational, prospective, longitudinal cohort study which will include patients, in a real-life setting, who are hospitalized for acute coronary syndrome (ACS) within 24 hours of symptom onset and who have a final diagnosis of Unstable Angina (UA), ST-Elevation Myocardial Infarction (STEMI) or Non-ST-Elevation Myocardial Infarction (NSTEMI). Patients will undergo clinical assessments and receive the standard medical care as determined by the treating cardiologist. Patients will not receive experimental intervention or experimental treatment as a consequence of their participation in the EPICOR-RUS observational study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older of either gender or race
* Diagnosis of STEMI, NSTEMI or UA confirmed using the following definitions

Exclusion Criteria:

* UA, STEMI and NSTEMI precipitated by or as a complication of surgery, trauma, or gastrointestinal (GI) bleeding or post-Percutaneous coronary intervention (PCI).
* UA, STEMI and NSTEMI occurring in patients already hospitalized for other reasons.
* Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient (e.g. tourist, non-native speaker or does not understand the local language, psychiatric disturbances).
* Already included in the EPICOR-RUS study.
* Presence of serious/severe co-morbidities in the opinion of the investigator which may limit short term (i.e. 6 month) life expectancy.
* Current participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical Practice
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Short- and long-term medication and treatment prescribed by physicians in real-life setting | up to 2 years

SECONDARY OUTCOMES:
clinical outcome (Cardiovascular events) | up to 2 years
quality of life (EQ-5D questionnaire) | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Stepanov, Study Director — AstraZeneca; Mikhail Ruda, Principal Investigator — RKNPK
Locations (19):
- Russia (19):
  - Research Site, Barnaul
  - Research Site, Cheboksary
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Kirov
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, N.Novgorod
  - Research Site, Novosibirsk
  - Research Site, Petrozavodsk
  - Research Site, Rostov-on-Don
  - Research Site, S-Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research site, Tomsk
  - Research Site, Tyumen
  - Research Site, Yekaterinburg

REFERENCES:
- [Derived] Ruda MY, Averkov OV, Khomitskaya YV. Long-term follow-up of antithrombotic management patterns in patients with acute coronary syndrome in Russia: an observational study (EPICOR-RUS study). Curr Med Res Opin. 2017 Jul;33(7):1269-1276. doi: 10.1080/03007995.2017.1313214. Epub 2017 Apr 19. PMID 28420281